CLINICAL TRIAL: NCT03762369
Title: Multi Center, Randomized, Double-blind, Active Controlled, Parallel Design, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-351 in Primary Open Angle Glaucoma or Ocular Hypertension Patients
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of CKD-351
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 171GLC18006
Record Dates: First submitted 2018-11-14; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension
Keywords: Primary Open-angle Glaucoma; Ocular Hypertension; CKD-351
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CKD-351 (Experimental): Latanoprost+D930
  Interventions: Drug: CKD-351; Drug: D930
- Latanoprost (Active Comparator)
  Interventions: Drug: Latanoprost; Drug: Placebo of CKD-351; Drug: Placebo of D930
- D930 (Active Comparator)
  Interventions: Drug: D930; Drug: Placebo of CKD-351

INTERVENTIONS:
Drug: CKD-351 — twice a day
  Other Names: Latanoprost+D930
  Arms: CKD-351
Drug: Latanoprost — once a day
  Arms: Latanoprost
Drug: D930 — three times a day
  Arms: CKD-351; D930
Drug: Placebo of CKD-351 — once a day
  Arms: Latanoprost
Drug: Placebo of CKD-351 — twice a day
  Arms: D930
Drug: Placebo of D930 — three times a day
  Arms: Latanoprost

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of CKD-351.

DETAILED DESCRIPTION:
Multi center, Randomized, Double-blind, Active controlled, Parallel design, Phase 3 trial to evaluate the efficacy and safety of CKD-351 in primary open angle glaucoma or ocular hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

1. More than the age of 19 years old
2. Subjects who has primary Open-Angle Glaucoma or Ocular Hypertension
3. Subjects who sign on an informed consent form willingly

Exclusion Criteria:

1. Subjects with IOP(Intraocular Pressure) ≥35 mmHg at Visit 1 and Visit 2 (AM 09:00) at more than one eye
2. Subjects with a maximum corrected visual acuity ≤ 0.3 in the selected evaluation eye at Visit 2
3. Subjects who were diagnosed as below with monocular or both eye

   * Acute or Chronic Closed-Angle Glaucoma
   * Secondary Glaucoma
   * Pseudoexfoliation Glaucoma
   * Neovascular Glaucoma
   * Aphakia
   * Phacocyst capsular torn intraocular lens
4. Subjects with significant eye symptoms/signs(Abscesses, diplopia) or severe visual field impairment(Mean Deviation ≥ -25dB)
5. Subjects with severe dry eye syndrome or progressive retinal disease(Retinal degeneration, Diabetic retinopathy, Retinal detachment, Macular edema)
6. Subjects with inflammatory/infectious eye disease and active eye disease within the last 3 months
7. Subjects who have medical history following

   * Subjects with significant history of ocular trauma during the last 6 months, or who underwent surgical ophthalmic surgery
   * Subjects who received topical or systemic steroids within the last 1 months
8. Subjects who wore need to wear contact lenses during the study
9. Women who are nursing, pregnant or planning pregnancy during the study
10. Subjects with bronchial asthma or history
11. Subjects with severe renal impairment (creatinine clearance <30 ml / min at screening) or hyperchloremic acidosis
12. Subjects who have received any other investigational product within 1 month prior to randomization
13. Impossible subjects who participate in clinical trial by investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2018-12-07 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean intraocular pressure at 12 weeks compared to baseline | Baseline, 12 weeks

SECONDARY OUTCOMES:
Change in mean intraocular pressure at 4 weeks, 8weeks compared to baseline | Baseline, 4 weeks, 8 weeks
Changes in intraocular pressure by measurement time | 4 weeks, 8 weeks, 12 weeks
  IOP variation by measurement time

OTHER OUTCOMES:
Safety assessed by number of participants with treatment-related adverse events | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: KiHo Park, Principal Investigator — Seoul National University Hosipital
Locations (1):
- Seoul National University Hosipital, Seoul, Jongno, South Korea

IPD SHARING:
Plan to Share IPD: No